CLINICAL TRIAL: NCT04041726
Title: Intraoperative Spillage of Bile and Gallstones During Laparoscopic Cholecysetectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar mohamed ahmed mohamed, Resident at general surgery department, Assiut University
Other Study IDs: Bile spillage intraoperative
Record Dates: First submitted 2019-07-27; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Cholecystitis; Gallstone
MeSH Terms: conditions — Cholecystitis; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. determine the most important factors which is responsible for the outcome post bile and gallstones spillage during laparoscopic cholecystectomy
2. the management of complications of bile and gallstones spillage

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is preferred surgical treatment for symptomatic gallstones .laparscopic procedure is superior to open procedue .the incidence of gallbladder perforation and spillage of bile and gallstones has been found as high as 40% .complications and management of gall bladder perforation and spillage of gallstones and bile

ELIGIBILITY:
Inclusion Criteria:

* all age groups
* only laparoscopic cholecystectomy
* all types ,numbers and sizes os gall stones

Exclusion Criteria:

* open cholecystectomh
* patient refuse to enrol this study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Results from intraoperative spillage of bile and gallstones intra abdomen during laparascopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Our purpose was to report the occurrence of complications following spilled gallstones during laparoscopic cholecystectomy at assiut university Hospital | Follow up complication for 6 months postoperative by abdominal ultrasound and multiple slice ct abdomen if needed
  Complications of intraoperative spilled gallstones and bile in laparoscopic cholecystectomy (inta abdominal abscess and localized bile collection ) and follow up for late complications